CLINICAL TRIAL: NCT06749392
Title: An Individual-specific Understanding of How Synchrony Becomes Curative
Brief Title: An Individual-specific Synchrony Signature
Acronym: SynSig
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Responsible Party: Principal Investigator, Sigal Zilcha Mano, Full professor, University of Haifa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 101123661
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Major Depressive Disorder
Keywords: Synchrony; Therapeutic relationship; Trait-like; State-like; Multi-modal; Mechanisms of change
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supportive-expressive psychotherapy (Experimental): Participants will receive supportive-expressive therapy for depressive disorder for 16 weeks.
  Interventions: Behavioral: Supportive-expressive treatment
- Waiting list (No Intervention): Participants will wait for treatment for 16 weeks. After the waiting the participants will receive in a supportive-expressive treatment for depressive disorder for 16 weeks.

INTERVENTIONS:
Behavioral: Supportive-expressive treatment — Sixteen weeks of a time-limited psychodynamic therapy adapted for depression that includes the use of expressive techniques, such as interpretation, confrontation, clarification and the use of supportive techniques, such as affirmation and empathic validation. This treatment postulates insight as its core mechanism of change.
  Arms: Supportive-expressive psychotherapy

SUMMARY:
This study aims to establish synchrony as an individual-specific mechanism of therapeutic change and offers novel insights into the mechanisms of curative interpersonal processes. The study identifies individual-specific trait-like synchrony signature and investigates the associations between synchrony signature, the individual's trait-like characteristics, and mental health, among participants diagnosed with Major Depressive Disorder. The study further investigates how deterministic the trait-like synchrony signature is by identifying for whom, how, and when changes are anticipated. Additionally, it examines whether synchrony signature transfers to relationships with the therapist, whether and how it changes throughout treatment, and whether such potential changes are associated with improvements in mental health. Synchrony is recognized as a key driver of collaborative, affiliative, and curative relationships. While its potential role in improving mental health through interpersonal relationships has sparked growing interest, particularly in psychotherapy, the field is at a crossroads, with mixed findings challenging the widespread theoretical assumption that "more synchrony is better." This study introduces a personalized framework that emphasizes individual-specific synchrony signatures, shifting from generalized assumptions to tailored understanding and interventions. The study explores how synchrony can transform relationships into curative ones by leveraging individual-tailored changes in synchrony signatures in psychotherapy. The potential impact is vast. Tailoring synchrony to individual-specific signatures represents a paradigm shift from a one-size-fits-all approach to personalized interventions. This personalized framework could revolutionize mental health care by facilitating the development of targeted strategies that enhance treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Current major depressive disorder based on the Diagnostic and Statistical Manual of Mental Disorders-5, and scores above 14 on the 17-item Hamilton rating scale for depression at two consecutive assessments, one week apart.
* For participants using psychiatric medication, the dosage must be stable for at least three months before the beginning of the study, and they will be asked to maintain stable dosage during the treatment
* Age between 18 and 65 years
* Hebrew language proficiency
* Provision of written informed consent.

Exclusion Criteria:

* Current risk of suicide or self-harm
* Current substance abuse disorders
* Current or past schizophrenia or psychosis, bipolar disorder, or severe eating disorder requiring medical monitoring
* History of organic mental disease
* Currently in psychotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-11-22 (Actual); Primary Completion 2030-03-30 (Estimated); Study Completion 2030-03-30 (Estimated)

PRIMARY OUTCOMES:
Weekly change in Hamilton rating scale for depression (HRSD) | Measured at baseline and every week for 16 weeks of treatment
  A 17-item clinically administered measure assessing the severity of depression. Each item is rated on a scale ranging from 0 (don't have) to 4 (sever) or 0 (don't have) to 2 (sever). The total score ranges between 0 and 52, where higher scores indicate worse outcome.

SECONDARY OUTCOMES:
Weekly change in Beck Depression Inventory (BDI) | Measured at baseline, every week for 16 weeks of treatment, then once a month for four months and follow up after a year.
  A 21-item, self-rated scale that evaluates key symptoms of depression. Each item is rated on a scale ranging from 0 (don't have) to 3 (sever). The total score ranges between 0 and 63, where higher scores indicate worse outcome.
Weekly change in Outcome Questionnaire (OQ) | Measured at baseline, every week for 16 weeks of treatment, then once a month for four months and follow up after a year.
  A 30 items self-report measure designed to assess patient therapy outcomes on three primary dimensions: (a) subjective discomfort, (b) interpersonal relationships, and (c) social role performance. Each item is rated on a scale ranging from 0 (never) to 4 (almost always). The total score ranges between 0 and 120, where higher scores indicate worse outcome.
Trajectories of change in Quality of Life Enjoyment and Satisfaction- Short Version (Q-LES-Q) | Measured at baseline, six times during the treatment (weeks 1, 2, 4, 8, 12, 16), then once a month for four months and follow up after a year.
  A 16-item self report measure designed to assess quality of life enjoyment and satisfaction. Each item is rated on a scale ranging from 1 (not at all) to 5 (extremely). The total score ranges between 16 and 80, where higher scores indicate better outcome.
Experiences in Close Relationships Questionnaire (ECR) | Measured at baseline, six times during the treatment (weeks 1, 2, 4, 8, 12, 16), then once a month for four months and follow up after a year.
  A 36-item self-report measure designed to assess adult attachment styles. The measurement data will be aggregated into two sub-scales: anxiety and avoidance. Each item is rated on a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). The total score on each subscale ranges between 18 and 126, where higher scores indicate worse outcome.
Trajectories of change in Inventory of Interpersonal Problems (IIP-32) | Measured at baseline, six times during the treatment (weeks 1, 2, 4, 8, 12, 16), then once a month for four months and follow up after a year.
  A 32-item self-report measure designed to assess interpersonal problems. Each item is rated in terms of how distressing the problem is for the individual on a scale ranging from 0 (not at all) to 4 (extremely). The total score ranges between 0 and 128, where higher scores indicate higher interpersonal problems, worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Haifa, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No
Data will not be shared due to ethical reasons.

REFERENCES:
- [Derived] Zilcha-Mano S, Bouknik Y, Malka M, Krasovsky T. An individual-specific understanding of how synchrony becomes curative: study protocol. BMC Psychiatry. 2025 Jun 6;25(1):587. doi: 10.1186/s12888-025-06539-3. PMID 40481468